CLINICAL TRIAL: NCT05121259
Title: Feasibility and Acceptability of an Online Web-based Physical Activity Program, for Those Living With and Beyond Lung Cancer.
Brief Title: Feasibility and Acceptability of an Web-based Physical Activity Program, for Those Diagnosed With Lung Cancer.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hull (Other)
Collaborators: Hull University Teaching Hospitals NHS Trust (Other Government)
Responsible Party: Principal Investigator, Cynthia Forbes, Career Development Fellow, University of Hull
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RS145-281450-JC
Record Dates: First submitted 2021-10-20; First posted 2021-11-16 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Lung Cancer; Survivorship
Keywords: Physical Activity; Exercise; Digtial Technology
MeSH Terms: conditions — Lung Neoplasms; Motor Activity

STUDY DESIGN:
Intervention Model Description: Single group feasibility study. Upon obtaining informed consent, participants will be allocated to the intervention group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise Guide (Experimental): Single group feasibility group. Single group (intervention group) will be given access to the intervention (Exercise Guide UK) for eight-weeks.
  Interventions: Other: ExerciseGuide Intervention Group

INTERVENTIONS:
Other: ExerciseGuide Intervention Group — The single group which will be given access to the eight-week ExerciseGuide UK website containing a tailored physical activity programme and supportive and educational resources.

SUMMARY:
Lung cancer is a life changing disease which can cause negative effects on an individual's ability to perform daily tasks and their quality of life (QoL). Lung cancer is the third most common cancer in the UK and is estimated affects approximately 33,000 individuals per year.

The most common side effects from lung cancer and treatments are breathlessness, fatigue, nausea, diarrhoea, and depression. Those living beyond cancer often suffer from extreme feelings of isolation and have increased chance of cardiovascular disease and diabetes.

Physical activity is a vital component of the prevention and management of cancer. Being active can improve one's physical health (ability to carry out tasks of daily living and breathlessness) and emotional wellbeing (feelings of depression and isolation).

Electronic platforms (websites and mobile applications) are increasingly popular within developing nations, particularly with products that aim to increase and keep track of physical activity. Though, literature suggests older adults prefer websites opposed to mobile applications. Online delivery of physical activity could be highly beneficial for patients living with and beyond cancer, reducing the location-based inequality of those who can not attend face-to-face programmes, allowing individuals to carry out a session whenever they can, in the comfort of their own home.

Exploring how those living with and beyond lung cancer use a website and investigating the feasibility and acceptability on an online platform which aims to provide tailored physical activity programs will provide fundamental data and possible supporting data for a randomised controlled trail (RCT).

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years of age or older.
* Have had a lung cancer diagnosis.
* Be able to speak and read in English.
* Willing and able to provide informed consent.
* Have internet connectivity.
* Access to a laptop, computer, or smart device to access the web-based platform.

Exclusion Criteria:

* Psychological or linguistic inability to provide informed consent.
* Physical or psychological impairments which prevent or inhibit participation in physical activity. Examples include:

  * Uncontrolled atrial fibrillation
  * Abdominal aortic aneurysm (AAA)
  * Recent heart attack (less than one year)
  * Recent stroke (less than one year)
  * Psychiatric disorder
  * Those who lack capacity under the Mental Capacity Act 2005 (MCA).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-11-22 (Actual); Primary Completion 2022-08-08 (Actual); Study Completion 2022-08-11 (Actual)

PRIMARY OUTCOMES:
The recruitment rate (Website Feasibility) | 39 weeks
  The recruitment rate will be established by the number of potential participants approached and how many agree to participate.
  The recruitment rate will be provided in a factorial or percentage format.
The retention rate (Website Feasibility) | 39 weeks
  The retention rate will be given based on the initial value of those who provide consent vs those who complete the eight-week intervention.
  The retention rate will be provided in a factorial or percentage format.
Participant Satisfaction (Acceptability) | 39 weeks
  The metric which will be assessed to explore acceptability will be satisfaction.
  Satisfaction will be explored in four approaches:
  1. Satisfaction via research team developed questionnaire. The questionnaire will be a five-point Likert scale reporting method from "Strongly Agree" to "Strongly Disagree" in relation to their agreement to statements.
  2. Real-time open-ended feedback will be collected upon the first completion of a module
  3. Systems Usability Scale (Brooke, 1986). The 10-item questionnaire will provide a five-point Likert scale reporting method from "Strongly Agree" to "Strongly Disagree" in relation to their agreement to statements.
  4. A selection of participants based on recruitment will be asked to take part in an interview to further explore satisfaction and acceptability. An interview guide covering the experience of using the website, concerns, and suggested revisions will be followed. The interviews will be transcribed verbatim and analysed.

SECONDARY OUTCOMES:
Quality of Life (or Global Health Status) will be assessed using the EORTC QLQ-C30 (version 3). | Eight weeks
  Quality of Life (or Global Health Status) will be assessed using the EORTC QLQ-C30 (version 3). The scoring value will be provided as a numerical value from the questionnaire and compared at baseline and study completion.
  The questionnaire used a four-point Likert scale reporting method 1, "Not at all"; 2, "A Little"; 3, "Quite a bit"; and 4, "Very much" in relation to their agreement to statements. Two questions (Q29 ad Q30) use a seven-point Likert scale reporting method ranging from 1 (Very poor) to 7 (Excellent).
Fatigue will be assessed using the EORTC QLQ-C30 (version 3 | Eight weeks
  Fatigue will be assessed using the EORTC QLQ-C30 (version 3). The scoring value will be provided in a numerical value from the questionnaire and compared at baseline and study completion.
  The questionnaire used a four-point Likert scale reporting method 1, "Not at all"; 2, "A Little"; 3, "Quite a bit"; and 4, "Very much" in relation to their agreement to statements.
Pain will be assessed using the EORTC QLQ-C30 (version 3) | Eight weeks
  Pain will be assessed using the EORTC QLQ-C30 (version 3). The scoring value will be provided in a numerical value from the questionnaire and compared at baseline and study completion.
  The questionnaire used a four-point Likert scale reporting method 1, "Not at all"; 2, "A Little"; 3, "Quite a bit"; and 4, "Very much" in relation to their agreement to statements.
Breathlessness | Eight weeks
  Breathlessness will be assessed using the EORTC QLQ-C30 (version 3). The scoring value will be provided in a numerical value from the questionnaire and compared at baseline and study completion.
  The questionnaire used a four-point Likert scale reporting method 1, "Not at all"; 2, "A Little"; 3, "Quite a bit"; and 4, "Very much" in relation to their agreement to statements.
Physical Functioning | Eight weeks
  Physical functioning will be assessed using the EORTC QLQ-C30 (version 3). The scoring value will be provided in a numerical value from the questionnaire and compared at baseline and study completion.
  The questionnaire used a four-point Likert scale reporting method 1, "Not at all"; 2, "A Little"; 3, "Quite a bit"; and 4, "Very much" in relation to their agreement to statements.
Emotional Functioning | Eight weeks
  Emotional functioning will be assessed using the EORTC QLQ-C30 (version 3). The scoring value will be provided in a numerical value from the questionnaire and compared at baseline and study completion.
Hospital Anxiety Depression Scale (HADS) | Eight weeks
  Hospital Anxiety Depression Scale (HADS) will be used pre-and post-study to explore changes in anxiety and depression.
  The HADS assigns statements to a numerical value (between 0 and 3) which is selected in agreement to the statement. These scores are totalled providing an overall score for both Anxeity and Depression.

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia C Forbes, PhD, Study Chair — University of Hull
Locations (1):
- Queen's Centre for Oncology and Haematology (Castle Hill), Hull, East Riding Of Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will be retained and stored for five years within an online secure folder within the Hull York Medical School server. Post five years, the data will be permanently destroyed by IT services based at the University of Hull. Per the data management plan, data will be anonymised and presented in publications arising from this study, including but no limited to the doctoral thesis of Mr. Jordan Curry and scientific article publications.
  Only Dr Forbes and Mr Curry will have access to the full IPD. In the thesis, blank documents pertaining to this study (informed consent form, information document, etc), will be provided.

REFERENCES:
- [Derived] Curry J, Lind M, Short CE, Vandelanotte C, Evans HEL, Pearson M, Forbes CC. Evaluating a web-based computer-tailored physical activity intervention for those living with and beyond lung cancer (ExerciseGuide UK): protocol for a single group feasibility and acceptability study. Pilot Feasibility Stud. 2022 Aug 13;8(1):182. doi: 10.1186/s40814-022-01129-6. PMID 35964141